CLINICAL TRIAL: NCT00332904
Title: Effect of Betablocker or Aldosterone Antagonist Therapy on Oxygenation, Peripheral and Cardiac Hemodynamics and Humoral Systems
Brief Title: Effect of Betablocker or Aldosterone Antagonist Therapy on Patients With Liver Cirrhosis
Acronym: PEKASYS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Christine Duemcke, MD, Hvidovre Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD-0606-HH-UH-DK
Record Dates: First submitted 2006-05-31; First posted 2006-06-02 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-06

CONDITIONS: Liver Cirrhosis; Portal Hypertension
Keywords: betablocker; aldosterone antagonist; peripheral haemodynamics; cardiac haemodynamics; oxygenation
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal | interventions — Propranolol; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- beta (Active Comparator): patients with liver cirrhosis, treated with betablocker
  Interventions: Drug: propranolol
- spiron (Active Comparator): patients with liver cirrhosis, treated with aldosterone antagonist
  Interventions: Drug: spironolactone
- control (No Intervention): patients with liver cirrhosis, no treatment

INTERVENTIONS:
Drug: propranolol — tablet 80 mg pr. day in a period of 3 weeks, evt. dose adjustment
  Arms: beta
Drug: spironolactone — tablet 200 mg pr. day in 3 weeks, evt. dose adjustment
  Arms: spiron

SUMMARY:
The study´s purpose is to investigate the effect of beta blockade or aldosterone antagonist therapy on oxygenation, peripheral and cardiac hemodynamics and humoral systems, in patients with liver cirrhosis.

DETAILED DESCRIPTION:
Cardio-pulmonal complications to patients with liver cirrhosis and portal hypertension determine the patients' prognosis. Most patients have hemodynamical changes in circulation with increased cardiac output and decreased systolic function in stress. Endothelial dysfunction is a parameter for bad prognosis in cardiovascular disease. The Renin-angiotensin-aldosterone-system plays an important role in natrium and volume regulation. Descriptions of changes in the peripheral circulation and oxygenation have been deficient up to now.

Patients with liver cirrhosis and portal hypertension are betablockers and/or aldosterone antagonists routine treatment - effects on peripheral hemodynamics and oxygenation in relation to central hemodynamic changes are deficient.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis
* Clinical indication for treatment with betablocker or aldosterone antagonist
* Must not have been treated earlier with betablocker or aldosterone antagonist
* Must have been alcohol abstinent for more than 4 weeks

Exclusion Criteria:

* Gastrointestinal bleeding in the last 2 weeks
* Encephalopathy > grade 1
* Acute medical conditions
* Malignant disease
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-08; Primary Completion 2008-07 (Actual); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
effect of treatment on hemodynamic and cardiac parameters | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Soeren Moeller, MD, DMSc, Study Director — Hvidovre University Hospital
Locations (1):
- Department of Clinical Physiology and Nuclear Medicine, and Department for Gastrointestinal Medicine, Hvidovre Hospital, Hvidovre, Denmark